CLINICAL TRIAL: NCT01650701
Title: A PHASE 3 OPEN-LABEL RANDOMIZED STUDY TO COMPARE THE EFFICACY AND SAFETY OF RITUXIMAB PLUS LENALIDOMIDE (CC-5013) VERSUS RITUXIMAB PLUS CHEMOTHERAPY FOLLOWED BY RITUXIMAB IN SUBJECTS WITH PREVIOUSLY UNTREATED FOLLICULAR LYMPHOMA The "RELEVANCE" Trial (Rituximab Lenalidomide Versus ANy ChEmotherapy)is Being Conducted as Two Companion Studies: RV-FOL-GELARC-0683 (N=750) and RV-FOL-GELARC-0683C (N=250); the Combined Total of 1000 Patients Enrolled in Both Studies Will be Analyzed.
Brief Title: A Phase 3 Open Label Randomized Study to Compare the Efficacy and Safety of Rituximab Plus Lenalidomide (CC-5013) Versus Rituximab Plus Chemotherapy Followed by Rituximab in Subjects With Previously Untreated Follicular Lymphoma
Acronym: RELEVANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-FOL-GELARC-0683; 2011-002792-42 (EudraCT Number)
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; non-hodgkins follicular lymphoma; treatment for follicular lymphoma; rituximab treatment; rituximab and lenalidomide treatment
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenalidomide + Rituximab (Experimental): * Lenalidomide dose 20-mg on days 2-22 every 28 days x 6 cycles, if CR then 10-mg on days 2-22 every 28 days for 12 cycles. PR after 6 cycles, continue 20 mg for 3~6 cycles and then 10 mg on days 2-22 every 28-day cycles for upto 18 cycles
  * Rituximab, 375 mg/m2 on days 1, 8, 15 and 22 of cycle 1, day 1 of cycles 2 to 6; 8 weeks later responding patients continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Interventions: Drug: Rituximab; Drug: Lenalidomide
- Control (Active Comparator): • ONE of the following: Rituximab - CHOP, Rituximab - CVP, Rituximab - Bendamustine. 7 to 8 weeks later responding patients will continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Interventions: Drug: Rituximab - CHOP; Drug: Rituximab - CVP; Drug: Rituximab - Bendamustine

INTERVENTIONS:
Drug: Rituximab — • Rituximab, 375 mg/m2 on days 1, 8, 15 and 22 of cycle 1, day 1 of cycles 2 to 6; 8 weeks later responding patients continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Other Names: mabthera; rituxan
  Arms: Lenalidomide + Rituximab
Drug: Lenalidomide — • Lenalidomide dose 20-mg on days 2-22 every 28 days x 6 cycles, if CR then 10-mg on days 2-22 every 28 days for 12 cycles. PR after 6 cycles, continue 20 mg for 3~6 cycles and then 10 mg on days 2-22 every 28-day cycles for upto 18 cycles
  Other Names: Revlimid
  Arms: Lenalidomide + Rituximab
Drug: Rituximab - CHOP — six cycles of R-CHOP in 21 day cycles followed by two 21 day cycles of 375 mg/m2 rituximab; and 7 weeks later responding patients continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles
  Arms: Control
Drug: Rituximab - CVP — eight cycles of R-CVP in 21 day cycles; and 7 weeks later responding patients continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles,
  Arms: Control
Drug: Rituximab - Bendamustine — six cycles of R-B in 28 day cycles and 8 weeks later responding patients continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Arms: Control

SUMMARY:
The purpose of this study is to find out if lenalidomide when given along with rituximab can help to control the disease and also increase the length of your response (complete or partial response) compared to the standard of care rituximab chemotherapy treatment.

DETAILED DESCRIPTION:
Follicular Lymphoma (FL) is a cancer of a B lymphocyte, a type of white blood cell. FL is typically a slowly progressing but incurable disease. Follicular lymphoma cells produce a specific defect in the patient's immune system impairing their ability to control their cancer. Lenalidomide has been shown to reverse the specific immune defect caused by FL in the patient. By including lenalidomide, the RELEVANCE study aims to eliminate the cancer while restoring the patient's immune competence.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20+ follicular lymphoma grade 1, 2 or 3a
* Have no prior systemic treatment for lymphoma.
* Must be in need of treatment
* Bi-dimensionally measurable disease with at least one mass lesion > 2 cm that was not previously irradiated.
* Stage II, III or IV disease.
* Must be ≥ 18 years and sign an informed consent.
* Performance status ≤ 2 on the ECOG scale.
* Adequate hematological function (unless abnormalities are related to lymphoma infiltration of the bone marrow)
* Willing to follow pregnancy precautions

Exclusion Criteria:

* Clinical evidence of transformed lymphoma by investigator assessment or Grade 3b follicular lymphoma.
* Patients taking corticosteroids during the last 4 weeks, unless administered at a dose equivalent to < 10 mg/day prednisone (over these 4 weeks).
* Major surgery (excluding lymph node biopsy) within 28 days prior to signing informed consent.
* Known Seropositive for or active viral infection with hepatitis B virus (HBV), hepatitis C virus (HCV)or human immunodeficiency virus (HIV).
* Life expectancy < 6 months.
* Known sensitivity or allergy to murine products.
* Prior history of malignancies, other than follicular lymphoma, unless the patient has been free of the disease for ≥ 10 years.
* Prior use of lenalidomide.
* Neuropathy > Grade 1.
* Presence or history of CNS involvement by lymphoma.
* Patients who are at a high risk for a thromboembolic event and are not willing to take venous thromboembolic (VTE) prophylaxis.
* serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) > 3x upper limit of normal (ULN), except in patients with documented liver or pancreatic involvement by lymphoma
* total bilirubin > 2.0 mg/dl (34 µmol/L) except in cases of Gilberts Syndrome and documented liver involvement by lymphoma
* creatinine clearance of < 30 mL/min
* Pregnant or lactating females.
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study, or which confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
COMPLETE RESPONSE RATE | Timeframe: CR/CRu rate at 120 weeks
  Complete response (CR/CRu) rate at 120 weeks Response evaluation was as defined by International Working Group (IWG) Response Criteria (Cheson 1999). Complete response (CR) is defined as the complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms if present before therapy.
Progression Free Survival (PFS) | up to 13 years
  PFS is defined as the time from the start of study drug therapy to the 1st observation of disease progression or death due to any cause.

SECONDARY OUTCOMES:
Number of participants with adverse events | up to13 years
Time to Treatment Failure (TTF) | up to13 years
Event Free Survival (EFS) | up to13 years
Time to Next Anti-Lymphoma Treatment (TTNLT), | up to13 years
Time to Next Chemotherapy Treatment (TTNCT) | up to13 years
Overall Survival (OS) | up to13 years
Overall response rate at 120 weeks by International Working Group (IWG) 1999 criteria | up to13 years
Health related quality of life as measured by the EORTC QLQ-C30 | up to13 years

CONTACTS AND LOCATIONS:
Overall Officials: Franck Morschhauser, MD, PhD, Study Chair — The Lymphoma Study Association (LYSA)
Locations (35):
- Australia (3):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
- CHU Mont-Godinne, Yvoir, Belgium
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corp - Saint John Regional Hospital, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - UHN-Princess Margaret Hospital, Toronto, Ontario
  - CHUM Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Hôpital de l'Enfant-Jesus, CHU de Quebec, Québec, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- CHU Claude Huriez, Lille, France
- Germany (3):
  - Medizinische Klinik der Universität Tübingen, Tübingen, Baden-Wurttemberg
  - Uniklinik Köln, Cologne, Nordrhein
  - LMU Munchën - Klinikum Grosshadern, München
- Italy (2):
  - Sant'Andrea Hospital, Rome, Lazio
  - Policlinico Sant'Orsola-Malpighi, Bologna
- Instituto Português Oncologia, Lisbon, Portugal
- Spain (12):
  - Hospital Virgen del Rocio, Seville, Andaloucia
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Son Llatzer, Palma, Mallorca
  - Hospital Clínico de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Institut Català d'Oncologia de Girona (ICO Girona), Girona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Costa del Sol, Marbella
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Claudel A, Cottereau AS, Bachy E, Itti E, Feugier P, Rossi C, Lemonnier F, Camus V, Daguindau N, Cartron G, Nicolas-Virelizier E, Mboumba DL, Cardoso C, Bommier C, Tessoulin B, Fruchart C, Gilbert A, Durot E, Fleck E, Pica GM, Zerazhi H, Guidez S, Cheminant M, Sarkozy C, Xerri L, Vercellino L, Trabelsi N, Gomes L, Portugues C, Viailly PJ, Delfau-Larue MH, Morschhauser F. Combined PET and ctDNA response as a predictor of POD24 for follicular lymphoma after first-line induction treatment. Blood. 2025 Aug 21;146(8):913-925. doi: 10.1182/blood.2024027727. PMID 40499012
- [Derived] Laurent C, Trisal P, Tesson B, Seth S, Beyou A, Roulland S, Lesne B, Van Acker N, Cerapio JP, Chartier L, Guille A, Stokes ME, Huang CC, Huet S, Gandhi AK, Morschhauser F, Xerri L. Follicular lymphoma comprises germinal center-like and memory-like molecular subtypes with prognostic significance. Blood. 2024 Dec 12;144(24):2503-2516. doi: 10.1182/blood.2024024496. PMID 39374535
- [Derived] Morschhauser F, Nastoupil L, Feugier P, Schiano de Colella JM, Tilly H, Palomba ML, Bachy E, Fruchart C, Libby EN, Casasnovas RO, Flinn IW, Haioun C, Maisonneuve H, Ysebaert L, Bartlett NL, Bouabdallah K, Brice P, Ribrag V, Le Gouill S, Daguindau N, Guidez S, Pica GM, Garcia-Sancho AM, Lopez-Guillermo A, Larouche JF, Ando K, Gomes da Silva M, Andre M, Kalung W, Sehn LH, Izutsu K, Cartron G, Gkasiamis A, Crowe R, Xerri L, Fowler NH, Salles G. Six-Year Results From RELEVANCE: Lenalidomide Plus Rituximab (R2) Versus Rituximab-Chemotherapy Followed by Rituximab Maintenance in Untreated Advanced Follicular Lymphoma. J Clin Oncol. 2022 Oct 1;40(28):3239-3245. doi: 10.1200/JCO.22.00843. Epub 2022 Aug 10. PMID 35947804
- [Derived] Delfau-Larue MH, Boulland ML, Beldi-Ferchiou A, Feugier P, Maisonneuve H, Casasnovas RO, Lemonnier F, Pica GM, Houot R, Ysebaert L, Tilly H, Eisenmann JC, Le Gouill S, Ribrag V, Godmer P, Glaisner S, Cartron G, Xerri L, Salles GA, Fest T, Morschhauser F. Lenalidomide/rituximab induces high molecular response in untreated follicular lymphoma: LYSA ancillary RELEVANCE study. Blood Adv. 2020 Aug 11;4(14):3217-3223. doi: 10.1182/bloodadvances.2020001955. PMID 32673385
- [Derived] Morschhauser F, Fowler NH, Feugier P, Bouabdallah R, Tilly H, Palomba ML, Fruchart C, Libby EN, Casasnovas RO, Flinn IW, Haioun C, Maisonneuve H, Ysebaert L, Bartlett NL, Bouabdallah K, Brice P, Ribrag V, Daguindau N, Le Gouill S, Pica GM, Martin Garcia-Sancho A, Lopez-Guillermo A, Larouche JF, Ando K, Gomes da Silva M, Andre M, Zachee P, Sehn LH, Tobinai K, Cartron G, Liu D, Wang J, Xerri L, Salles GA; RELEVANCE Trial Investigators. Rituximab plus Lenalidomide in Advanced Untreated Follicular Lymphoma. N Engl J Med. 2018 Sep 6;379(10):934-947. doi: 10.1056/NEJMoa1805104. PMID 30184451